CLINICAL TRIAL: NCT02263508
Title: A Phase 1b/3, Multicenter, Trial of Talimogene Laherparepvec in Combination With Pembrolizumab (MK-3475) for Treatment of Unresectable Stage IIIB to IVM1c Melanoma (MASTERKEY-265)
Brief Title: Pembrolizumab With Talimogene Laherparepvec or Placebo in Unresected Melanoma
Acronym: MASTERKEY-265
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20110265; 2014-000185-22 (EudraCT Number); KEYNOTE-034 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2014-09-26; First posted 2014-10-13 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Melanoma
Keywords: Talimogene Laherparepvec; pembrolizumab; KEYNOTE-034; MASTERKEY-265
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1b was an open-label, single-arm study. Phase 3 was a randomized, double-blind, placebo-controlled study design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b: Talimogene Laherparepvec + Pembrolizumab (Experimental): Participants received talimogene laherparepvec at an initial dose of up to 4 mL 10⁶ plaque-forming units (PFU)/mL by intralesional injection. Subsequent doses of talimogene laherparepvec at up to 4 mL of 10⁸ PFU/mL began 3 weeks after the first dose and were administered every 2 weeks until disappearance of injectable lesions, complete response (CR), confirmed disease progression (PD) per modified Immune-related Response Criteria (irRC), intolerance of study treatment, 24 months from the date of the first dose of pembrolizumab, or end of study, whichever occurred first. Participants also received 200 mg pembrolizumab administered intravenously every 2 weeks starting at the time of the third dose of talimogene laherparepvec (week 6) until confirmed PD per modified irRC, treatment intolerance, 24 months from the first dose, or end of study, whichever occurred first.
  Interventions: Drug: Talimogene Laherparepvec; Drug: Pembrolizumab
- Phase 3 : Placebo + Pembrolizumab (Placebo Comparator): Participants received up to 4 mL placebo to talimogene laherparepvec by intralesional injection on day 1 of week 0. Subsequent doses of placebo (up to 4 mL) began 3 weeks after the first dose and were administered every 2 weeks until the fifth injection (week 9), and then synchronously with pembrolizumab thereafter every 3 weeks until disappearance of injectable lesions, complete response per modified Immune-related Response Criteria simulating Response Evaluation Criteria in Solid Tumors (irRC-RECIST) (iCR), confirmed iPD per modified irRC-RECIST, intolerance of study treatment, 24 months from the date of the first dose of placebo, or end of study, whichever occurred first. Participants also received 200 mg pembrolizumab administered intravenously every 3 weeks starting on day 1 of week 0, until confirmed iPD per modified irRC-RECIST, treatment intolerance, 24 months from the first dose, or end of study, whichever occurred first.
  Interventions: Drug: Pembrolizumab; Drug: Placebo
- Phase 3: Talimogene Laherparepvec + Pembrolizumab (Experimental): Participants received talimogene laherparepvec at an initial dose of up to 4 mL 10⁶ PFU/mL by intralesional injection on day 1. Subsequent doses of talimogene laherparepvec at 10⁸ PFU/mL (up to 4 mL) began 3 weeks after the first dose and were administered every 2 weeks until the fifth injection of talimogene laherparepvec (week 9), and then synchronously with pembrolizumab thereafter every 3 weeks until disappearance of injectable lesions, iCR, confirmed iPD per modified irRC-RECIST, intolerance of study treatment, 24 months from the date of the first dose of talimogene laherparepvec, or end of study, whichever occurred first. Participants also received 200 mg pembrolizumab administered intravenously every 3 weeks starting on day 1 of week 0, until confirmed iPD per modified irRC-RECIST, treatment intolerance, 24 months from the first dose, or end of study, whichever occurred first.
  Interventions: Drug: Talimogene Laherparepvec; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene laherparepvec administered by intratumoral injection
  Other Names: IMLYGIC®; OncoVEX^GM-CSF; T-VEC
  Arms: Phase 1b: Talimogene Laherparepvec + Pembrolizumab; Phase 3: Talimogene Laherparepvec + Pembrolizumab
Drug: Pembrolizumab — Administered at a dose of 200 mg as an intravenous infusion over approximately 30 minutes.
  Other Names: MK-3475; Keytruda®
Drug: Placebo — Administered by intratumoral injection
  Arms: Phase 3 : Placebo + Pembrolizumab

SUMMARY:
The primary objectives of the Phase 1b part of the study are to evaluate the safety, as assessed by incidence of dose limiting toxicity (DLT), of talimogene laherparepvec in combination with pembrolizumab in adults with previously untreated, unresectable, stage IIIB to IVM1c melanoma.

The primary objective of Phase 3 are to evaluate the efficacy of talimogene laherparepvec with pembrolizumab versus placebo with pembrolizumab, as assessed by progression-free survival (PFS) (response evaluation by blinded independent central review using modified Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) and overall survival (OS).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years with histologically confirmed diagnosis of melanoma and stage IIIB to IVM1c for whom surgery is not recommended.
* Subjects must have measurable disease and be a candidate for intralesional therapy administration into cutaneous, subcutaneous, or nodal lesions.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, hepatic, renal, and coagulation function.
* Subjects with serine/threonine protein kinase B-Raf V600 (BRAFV600) wild-type tumors must not have received any prior systemic anticancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy given in a non-adjuvant setting for unresectable stage IIIB to IVM1c melanoma.
* Subjects with B-Raf V600 (BRAFV600) mutated tumors who have received prior BRAF inhibitor therapy either alone or in combination with mitogen-activated protein kinase kinase (MEK) inhibitor as their only prior systemic therapy are eligible.
* Subjects who received prior adjuvant therapy for melanoma will not be excluded (including, but not limited to, interferon, ipilimumab, limb infusion/perfusion, or use of investigational agents in the adjuvant setting) with the exception that prior adjuvant therapy with inhibitors of programmed cell death-1 (PD-1) or programmed cell death ligand 1 (PD-L1) is not allowed. However, if the subject received adjuvant therapy, the subject must have completed therapy at least 28 days prior to enrollment.
* Subjects must have a tumor sample that is adequate for PD-L1 assessment prior to randomization.

Key Exclusion Criteria:

* Subjects must not have clinically active cerebral metastases.
* Subjects must not have primary uveal or mucosal melanoma, history or evidence of melanoma associated with immunodeficiency states or history of other malignancy within the past 3 years.
* Subjects may not have been previously treated with talimogene laherparepvec, any other oncolytic virus, pembrolizumab, or any other inhibitor of PD-1, PD-L1, or PD-L2.
* Subjects must not have history or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, other symptomatic autoimmune disease, documented history of autoimmune disease or syndrome requiring systemic treatment in the past 2 years (ie, with use of disease modifying agents, steroids or immunosuppressive agents) except vitiligo or resolved childhood asthma/atopy, or evidence of clinically significant immunosuppression.
* Subjects must not have active herpetic skin lesions or prior complications of herpetic infection and must not require intermittent or chronic treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (143):
- United States (35):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Duarte, California
  - Research Site, Encinitas, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Riverside, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Fridley, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Germantown, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (11):
  - Research Site, North Sydney, New South Wales
  - Research Site, Waratah, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Southport, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Woodville South, South Australia
  - Research Site, Geelong, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Murdoch, Western Australia
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Liège
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (4):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
- Research Site, Helsinki, Finland
- France (10):
  - Research Site, Bordeaux
  - Research Site, Grenoble
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (14):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Tübingen
  - Research Site, Würzburg
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion - Crete
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Pécs
  - Research Site, Szeged
- Italy (5):
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Meldola FC
  - Research Site, Milan
  - Research Site, Siena
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Nijmegen
- Poland (9):
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Konin
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (3):
  - Research Site, Almada
  - Research Site, Lisbon
  - Research Site, Porto
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (5):
  - Research Site, Groenkloof, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Parktown, Gauteng
  - Research Site, Kraaifontein
  - Research Site, Pretoria
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Donostia / San Sebastian, Basque Country
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Pamplona, Navarre
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Switzerland (5):
  - Research Site, Bellinzona
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Zurich
- United Kingdom (9):
  - Research Site, Birmingham
  - Research Site, Guildford
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Preston
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Ribas A, Dummer R, Puzanov I, VanderWalde A, Andtbacka RHI, Michielin O, Olszanski AJ, Malvehy J, Cebon J, Fernandez E, Kirkwood JM, Gajewski TF, Chen L, Gorski KS, Anderson AA, Diede SJ, Lassman ME, Gansert J, Hodi FS, Long GV. Oncolytic Virotherapy Promotes Intratumoral T Cell Infiltration and Improves Anti-PD-1 Immunotherapy. Cell. 2017 Sep 7;170(6):1109-1119.e10. doi: 10.1016/j.cell.2017.08.027. PMID 28886381
- [Background] Dummer R, Hoeller C, Gruter IP, Michielin O. Combining talimogene laherparepvec with immunotherapies in melanoma and other solid tumors. Cancer Immunol Immunother. 2017 Jun;66(6):683-695. doi: 10.1007/s00262-017-1967-1. Epub 2017 Feb 25. PMID 28238174
- [Background] Chesney JA, Ribas A, Long GV, Kirkwood JM, Dummer R, Puzanov I, Hoeller C, Gajewski TF, Gutzmer R, Rutkowski P, Demidov L, Arenberger P, Shin SJ, Ferrucci PF, Haydon A, Hyngstrom J, van Thienen JV, Haferkamp S, Guilera JM, Rapoport BL, VanderWalde A, Diede SJ, Anderson JR, Treichel S, Chan EL, Bhatta S, Gansert J, Hodi FS, Gogas H. Randomized, Double-Blind, Placebo-Controlled, Global Phase III Trial of Talimogene Laherparepvec Combined With Pembrolizumab for Advanced Melanoma. J Clin Oncol. 2023 Jan 20;41(3):528-540. doi: 10.1200/JCO.22.00343. Epub 2022 Aug 23. PMID 35998300
- [Derived] Watanabe D, Goshima F. Oncolytic Virotherapy by HSV. Adv Exp Med Biol. 2018;1045:63-84. doi: 10.1007/978-981-10-7230-7_4. PMID 29896663
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 134 centers in Australia, Canada, Europe, South Africa, South Korea, and the United States.
  Phase 1b was an open-label, single-arm study and Phase 3 was a randomized, double-blind, placebo-controlled study.
Pre-assignment Details: In Phase 3 participants were randomized equally to 1 of 2 arms. Randomization was stratified by stage of disease: less advanced stages (IIIB, IIIC, and IVM1a) versus more advanced stages (IVM1b and IVM1c) and by prior serine/threonine protein kinase B-Raf (BRAF) inhibitor therapy (no prior BRAF inhibitor versus BRAF inhibitor with or without mitogen-activated extracellular signal-regulated kinase [MEK] inhibitor).
Groups:
- Phase 1b: Talimogene Laherparepvec + Pembrolizumab: Participants received talimogene laherparepvec at an initial dose of up to 4 mL 10⁶ plaque-forming units (PFU)/mL by intralesional injection on day 1 of week 1. Subsequent doses of talimogene laherparepvec at up to 4 mL of 10⁸ PFU/mL began 3 weeks after the first dose and were administered every 2 weeks until disappearance of injectable lesions, complete response (CR), confirmed disease progression (PD) per modified Immune-related Response Criteria (irRC), intolerance of study treatment, 24 months from the date of the first dose of pembrolizumab, or end of study, whichever occurred first. Participants also received 200 mg pembrolizumab administered intravenously every 2 weeks starting at the time of the third dose of talimogene laherparepvec (week 6) until confirmed PD per modified irRC, treatment intolerance, 24 months from the first dose, or end of study, whichever occurred first.
- Phase 3: Placebo + Pembrolizumab: Participants received up to 4 mL placebo to talimogene laherparepvec by intralesional injection on day 1 of week 0. Subsequent doses of placebo (up to 4 mL) began 3 weeks after the first dose and were administered every 2 weeks until the fifth injection (week 9), and then synchronously with pembrolizumab thereafter every 3 weeks until disappearance of injectable lesions, complete response per modified Immune-related Response Criteria simulating Response Evaluation Criteria in Solid Tumors (irRC-RECIST) (iCR), confirmed iPD per modified irRC-RECIST, intolerance of study treatment, 24 months from the date of the first dose of placebo, or end of study, whichever occurred first. Participants also received 200 mg pembrolizumab administered intravenously every 3 weeks starting on day 1 of week 0, until confirmed iPD per modified irRC-RECIST, treatment intolerance, 24 months from the first dose, or end of study, whichever occurred first.
Period: Overall Study
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Started | 21 | 346 | 346
Received Talimogene Laherparepvec/Placebo | 21 | 345 | 343
Received Pembrolizumab | 21 | 345 | 343
Completed | 0 | 0 | 0
Not Completed | 21 | 346 | 346
Not completed — Withdrawal by Subject | 1 | 23 | 17
Not completed — Sponsor Decision | 12 | 165 | 182
Not completed — Lost to Follow-up | 2 | 7 | 7
Not completed — Death | 6 | 151 | 140

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab | Total
Number analyzed (Participants) | 21 | 346 | 346 | 713
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (13.4) | 62.3 (14.5) | 63.1 (13.7) | 62.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 127 | 147 | 287
  Male | 8 | 219 | 199 | 426
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 9 | 13 | 22
  Not Hispanic or Latino | 21 | 337 | 331 | 689
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 7 | 11
  Black (or African American) | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 21 | 335 | 327 | 683
  Other | 0 | 6 | 10 | 16
Disease Stage per the American Joint Committee on Cancer (AJCC) 7th Edition [Count of Participants; unit: Participants] — Stage IIIB: Ulcerated lesion and 1 lymph node or 2-3 nodes with micrometastasis, or any-depth lesion with no ulceration, and 1 lymph node or 2-3 nodes with macrometastasis; Stage IIIC: Ulcerated lesion and 1 lymph node with macrometastasis; 2-3 nodes with macrometastasis or ≥4 metastatic lymph nodes, matted lymph nodes, or in-transit met(s)/satellite(s); Stage IV: M1a: Spread to skin, subcutaneous tissue, or lymph nodes; normal lactate dehydrogenase (LDH) level; M1b: Spread to lungs, normal LDH; M1c: Spread to all other visceral organs, normal LDH or any distant disease with elevated LDH.
  Participants
    Stage IIIB - IVM1a | 9 | 169 | 169 | 347
    Stage IVM1b/c | 12 | 177 | 177 | 366
Prior Serine/Threonine Protein Kinase B-Raf (BRAF) Inhibitor Therapy [Count of Participants; unit: Participants] — Population: Prior BRAF inhibitor therapy was not collected in Phase 1b
  Participants
    number analyzed (Participants) | 0 | 346 | 346 | 692
    Yes |  | 29 | 29 | 58
    No |  | 317 | 317 | 634
Programmed Cell Death-1 Ligand 1 (PD-L1) Status [Count of Participants; unit: Participants] — PD-L1 expression in tumor cells was assessed at a central laboratory using a clinical trial immunohistochemistry assay (22C3 antibody) and scored on a unique melanoma (MEL) scale of 0 to 5; a score ≥ 2 (membranous staining in ≥ 1% of cells within tumor nests, including neoplastic cells and intercalated and contiguous immune cells) was considered positive.
  Participants
    Positive | 17 | 218 | 231 | 466
    Not Positive | 4 | 128 | 115 | 247
BRAF V600 Mutation Status [Count of Participants; unit: Participants] — Mutation status of v-raf murine sarcoma viral oncogene homolog B1 (BRAF) gene was based on a gene mutation that results in an amino acid substitution from valine (V) to glutamic acid (E) at codon 600 (V600E) and/or a substitution from valine to lysine (K) (V600K).
  Participants
    Mutation | 4 | 116 | 124 | 244
    Mutation not present | 17 | 215 | 211 | 443
    Missing/unknown | 0 | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any toxicity related to study drug which met any of the following criteria based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0:
  * Grade 4 non-hematologic toxicity.
  * Grade 3 or higher pneumonitis.
  * Grade 3 non-hematologic toxicity lasting > 3 days despite optimal supportive care, excluding grade 3 fatigue.
  * Any grade 3 or higher non-hematologic laboratory value if medical intervention was required, or the abnormality lead to hospitalization, or the abnormality persisted for > 1 week.
  * Febrile neutropenia grade 3 or grade 4.
  * Thrombocytopenia < 25 x 10^9/L if associated with a bleeding event which does not result in hemodynamic instability but required an elective platelet infusion, or a life-threatening bleeding event which resulted in urgent intervention and admission to intensive care unit.
  * Grade 5 toxicity (ie, death).
  * Any other intolerable toxicity leading to permanent discontinuation of talimogene laherparepvec or pembrolizumab.
Time Frame: The DLT evaluation period was 6 weeks from the initial administration of pembrolizumab (week 6 to 12).
Population: The DLT analysis set included DLT-evaluable participants enrolled in Phase 1b who had the opportunity to be on treatment for at least 6 weeks from the initial dose of pembrolizumab and received at least 2 doses of talimogene laherparepvec and 2 doses of pembrolizumab in combination (ie, on the same day), or those who otherwise experienced a DLT within 6 weeks after starting the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
Participants | 0

2. Primary Outcome: Phase 3: Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) Assessed Using Modified RECIST 1.1
Description: PFS per modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 is defined as the interval from randomization to the earlier event of progressive disease (PD) per modified RECIST 1.1 or death from any cause.
  PD: Increase in size of target lesions from nadir by ≥ 20% and ≥ 5 mm absolute increase above nadir, or the appearance of a new lesion.
  Median PFS was calculated using the Kaplan-Meier method. Participants without an event were censored at their last evaluable tumor assessment if available; otherwise on their randomization date.
  The primary analysis of PFS was specified to be conducted when 407 PFS events had occurred (data cut-off date 02 March 2020).
Time Frame: From randomization until the data-cut-off date of 02 March 2020; median (range) time on follow-up was 25.5 (0.6, 44.7) months in the Placebo + Pembrolizumab arm and 25.6 (0.3, 45.8) months in the Talimogene Laherparepvec + Pembrolizumab arm.
Population: All participants randomized in Phase 3.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
months | 8.5 [5.72 to 13.54] | 14.3 [10.25 to 22.11]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Superiority; p = 0.13, Stratified log-rank test; Stratified by randomization factors (disease stage, prior BRAF inhibitor therapy) and baseline PD-L1 status; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.71 to 1.04] — Cox proportional hazards model stratified by randomization factors (disease stage, prior BRAF inhibitor therapy) and baseline PD-L1 status

3. Primary Outcome: Phase 3: Overall Survival
Description: Overall survival (OS) is defined as the interval from randomization to death from any cause.
  Median overall survival was calculated using the Kaplan-Meier method. Participants without an event were censored at their last known alive date.
Time Frame: From randomization until the end of study; median (range) time on follow-up was 34.8 (0.6, 58.3) months in the Placebo + Pembrolizumab arm and 36.8 (0.3, 58.4) months in the Talimogene Laherparepvec + Pembrolizumab arm.
Population: All participants randomized in Phase 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Superiority; p = 0.77, Stratified log-rank test; Stratified by randomization factors (disease stage, prior BRAF inhibitor therapy) and baseline PD-L1 status; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.21] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Phase 1b: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) using the modified Immune-related Response Criteria (irRC), by Investigator assessment.
  CR was defined as the disappearance of all lesions; PR was defined as a decrease in tumor area ≥ 50% relative to baseline, response must have been confirmed by a second, consecutive assessment at least 4 weeks apart.
  Radiographic imaging for assessment of lesions was performed using computed tomography (CT), positron emission tomography (PET), magnetic resonance imaging (MRI), or ultrasound. Clinical measurement of cutaneous, subcutaneous, and palpable nodal tumor lesions was conducted with calipers.
Time Frame: Tumor assessments were performed at week 6 (prior to initiation of pembrolizumab), week 18, and every 12 weeks thereafter until confirmed PD or start of new anticancer treatment; median (range) time on follow-up was 58.6 (1.4, 61.6) months.
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab.
  Participants with no post-baseline tumor assessments were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
percentage of participants | 61.9 [38.4 to 81.9]

5. Secondary Outcome: Phase 1b: Best Overall Response (BOR)
Description: Best overall response is defined as the best overall visit response in the following order: CR, PR, stable disease (SD), progressive disease (PD), or unevaluable (UE), based on investigator assessment using the modified irRC up to the start of any subsequent anti-cancer therapy.
  CR was defined as the disappearance of all lesions; PR was defined as a decrease in tumor area ≥ 50% relative to baseline; PD was defined as an increase in tumor area ≥ 25% relative to nadir; and SD was defined as any outcome not meeting the criteria for response or PD with ≥ 77 days elapsed after enrollment. Responses and PD must have been confirmed by a second, consecutive assessment at least 4 weeks apart.
Time Frame: as for outcome 4
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
Participants
  Complete Response (CR) | 9
  Partial Response (PR) | 4
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 6
  Unable to Evaluate (UE) | 1

6. Secondary Outcome: Phase 1b: Durable Response Rate (DRR)
Description: DRR is defined as the percentage of participants with a best overall response of CR or PR using the modified irRC per Investigator assessment with a duration of response of at least 6 months.
  CR was defined as the disappearance of all lesions; PR was defined as a decrease in tumor area ≥ 50% relative to baseline, response must have been confirmed by a second, consecutive assessment at least 4 weeks apart.
Time Frame: as for outcome 4
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
percentage of participants | 57.1 [34.0 to 78.2]

7. Secondary Outcome: Phase 1b: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time from the date of an initial response (CR or PR) that is subsequently confirmed to the earlier of confirmed PD or death. Participants who had not ended their response at the time of analysis were censored at their last evaluable tumor assessment before start of the first subsequent anticancer therapy.
  CR was defined as the disappearance of all lesions; PR was defined as a decrease in tumor area ≥ 50% relative to baseline; PD was defined as an increase in tumor area ≥ 25% relative to nadir. Response and PD must have been confirmed by a second, consecutive assessment at least 4 weeks apart.
Time Frame: as for outcome 4
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab with a CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 13
months | NA [NA to NA] — Could not be estimated due to the low number of events

8. Secondary Outcome: Phase 1b: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a best overall response of CR, PR, or SD using the modified irRC per Investigator assessment.
  CR was defined as the disappearance of all lesions; PR was defined as a decrease in tumor area ≥ 50% relative to baseline, response must have been confirmed by a second, consecutive assessment at least 4 weeks apart; and SD was defined as any outcome not meeting the criteria for response or PD with ≥ 84 days elapsed after enrollment.
Time Frame: as for outcome 4
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
percentage of participants | 66.7 [43.0 to 85.4]

9. Secondary Outcome: Phase 1b: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from first dose to the earlier event of confirmed PD per modified irRC or death from any cause. PFS was estimated using the Kaplan-Meier method. Participants without an event were censored at their last evaluable tumor assessment.
Time Frame: From first dose until the end of study; median (range) time on follow-up was 70.6 (1.4, 74.5) months.
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
months | NA [NA to NA] — Could not be estimated due to the low number of events

10. Secondary Outcome: Phase 1b: Overall Survival (OS)
Description: Overall survival is defined as the interval from first dose to death from any cause.
  OS was estimated using the Kaplan-Meier method. Participants without an event were censored at their last known alive date.
Time Frame: From first dose until the end of study; median (range) time on follow-up was 70.6 (1.4, 74.5) months.
Population: All participants enrolled in Phase 1b who received ≥ 1 dose of talimogene laherparepvec or pembrolizumab
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21
months | NA [NA to NA] — Could not be estimated due to the low number of events

11. Secondary Outcome: Phase 3: Complete Response Rate Assessed Using Modified irRC-RECIST (iCRR)
Description: Complete response rate per modified Immune-related Response Criteria (irRC) simulating RECIST 1.1 (irRC-RECIST) is defined as the percentage of participants with a best overall response of complete response assessed using the modified irRC-RECIST (iCR) evaluated by blinded independent central review.
  iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment at least 4 weeks after the criteria were first met. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Modifications to the irRC-RECIST 1.1 included an increase in the total number of target lesions and new measurable lesions to 10 with a maximum of 5 target lesions per organ, and target lesions must have been measurable by CT or MRI only.
Time Frame: Tumor assessments were performed every 12 weeks after initiation of treatment until confirmed PD or start of new anticancer treatment; median (range) time on follow-up was 30.6 (0.6, 53.0) months and 31.4 (0.3, 52.5) months in each group, respectively.
Population: All participants randomized in Phase 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 8.1 [5.22 to 10.97] | 14.5 [10.75 to 18.16]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.012, Regression, Logistic; Logistic regression stratified by randomization stratification factors (disease stage and prior BRAF inhibitor therapy) and the baseline PD-L1 status; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.15 to 3.07] — Adjusted odds ratio estimated using logistic regression with randomization stratification factors and baseline PD-L1 status

12. Secondary Outcome: Phase 3: Progression Free Survival Assessed Using Modified irRC-RECIST (iPFS)
Description: PFS per modified irRC-RECIST is defined as the interval from randomization to the earlier event of progressive disease assessed by modified irRC-RECIST (iPD) evaluated by blinded independent central review, or death from any cause.
  iPD: Increase in tumor burden ≥ 20% and at least 5 mm absolute increase relative to nadir (minimum recorded tumor burden) confirmed by a repeat, consecutive assessment at least 4 weeks after the initial detection.
  Median iPFS was calculated using the Kaplan-Meier method. Participants without an event were censored at their last evaluable tumor assessment if available; otherwise on their randomization date.
  The primary analysis of iPFS was specified to be conducted when 256 iPFS events had occurred (data cut-off date 29 September 2020).
Time Frame: From randomization until the data cut-off date of 29 September 2020; median time on follow-up was 30.6 (0.6, 53.0) months in the Placebo + Pembrolizumab arm and 31.4 (0.3, 52.5) months in the Talimogene Laherparepvec + Pembrolizumab arm.
Population: All participants randomized in Phase 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 3 : Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
months | 25.3 [17.68 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Phase 3 : Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.14, Stratified log-rank test; Stratified by randomization factors (disease stage, prior BRAF inhibitor therapy) and baseline PD-L1 status; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.82 to 1.34] — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Phase 3: Overall Survival Excluding Stage IVM1c Participants
Description: Overall survival is defined as the interval from randomization to death from any cause.
  Median OS was calculated using the Kaplan-Meier method. Participants without an event were censored at the last known alive date.
Time Frame: as for outcome 3
Population: Participants randomized in Phase 3 with stage IIIB to IVM1a/b.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 203 | 201
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.47, Stratified log-rank test; Stratified by randomization factors (disease stage, prior BRAF inhibitor therapy) and baseline PD-L1 status; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.63 to 1.24] — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Phase 3: Objective Response Rate Assessed Using Modified RECIST 1.1
Description: ORR is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) assessed using modified RECIST version 1.1, evaluated by blinded independent central review.
  CR was defined as the disappearance of all lesions except lymph node short axis < 10 mm; PR was defined as a ≥ 30% reduction in sum of diameters in target lesions. Confirmation of CR or PR was not required.
  Modifications to conventional RECIST 1.1 included the following: target lesions were measurable on CT or MRI; otherwise, they were considered as nontarget lesions. A maximum of 10 target lesions was allowed with up to 5 per organ.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3; Participants with no post-baseline tumor assessments were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 41.3 [36.14 to 46.52] | 48.6 [43.29 to 53.82]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.081, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.97 to 1.79] — [estimate comment as in outcome 11, analysis 1]

15. Secondary Outcome: Phase 3: Best Overall Response Assessed Using Modified RECIST 1.1
Description: BOR is defined as the best overall visit response up to and including the first overall visit response of PD in the following order: CR, PR, SD, non-CR/Non-PD (NN), PD or UE per modified RECIST 1.1, evaluated by BICR.
  CR: Disappearance of all lesions except lymph node short axis < 10 mm; PR: ≥ 30% reduction in sum of diameters in target lesions. Confirmation of CR or PR was not required; NN: Persistence of ≥ 1 non-target lesions and/or maintenance of tumor marker level above normal limits; SD: Neither sufficient shrinkage of target lesions to qualify for CR or PR nor sufficient increase to qualify for PD and ≥ 84 days from randomization; PD: Increase from nadir by ≥ 20% or ≥ 5 mm of target lesions or any new lesion; Missing: No postbaseline assessment, or assessments on or after the start of first subsequent anticancer therapy, including complete or partial removal/reduction of any target lesion which contained melanoma on pathology evaluation or pathology results were unknown.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
Participants
  Complete response (CR) | 40 | 62
  Partial response (PR) | 103 | 106
  Stable disease (SD) | 30 | 28
  Non-CR/Non-PD (NN) | 16 | 11
  Progressive disease (PD) | 120 | 106
  Unevaluable (UE) | 11 | 3
  Missing | 26 | 30

16. Secondary Outcome: Phase 3: Durable Response Rate (DRR) Assessed Using Modified RECIST 1.1
Description: DRR is defined as the percentage of participants with a CR or PR per modified RECIST 1.1 evaluated by blinded independent central review, with a duration of response of ≥ 6 months.
  CR was defined as the disappearance of all lesions except lymph node short axis < 10 mm; PR was defined as a ≥ 30% reduction in sum of diameters in target lesions. Confirmation of CR or PR was not required.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 34.1 [29.11 to 39.10] | 42.2 [36.99 to 47.40]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.039, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.02 to 1.90] — [estimate comment as in outcome 11, analysis 1]

17. Secondary Outcome: Phase 3: Duration of Response (DOR) Assessed Using Modified RECIST 1.1
Description: Duration of response (DOR) is defined as the time from the date of an initial response of CR or PR to the earlier of PD per modified RECIST 1.1, or death. Participants who had not ended their response at the time of analysis were censored at their last evaluable tumor assessment date before start of the first subsequent anticancer therapy.
  CR was defined as the disappearance of all lesions except lymph node short axis < 10 mm; PR was defined as a ≥ 30% reduction in sum of diameters in target lesions. Confirmation of CR or PR was not required. PD was defined as an increase from nadir by ≥ 20% or ≥ 5 mm absolute increase above nadir of target lesions or appearance of any new lesion.
Time Frame: as for outcome 12
Population: Participants randomized in Phase 3 with a CR or PR per modified RECIST.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 143 | 168
months | NA [NA to NA] — Could not be estimated due to the low number of events | 43.7 [NA to NA] — Could not be estimated due to the low number of events

18. Secondary Outcome: Phase 3: Disease Control Rate (DCR) Assessed Using RECIST 1.1
Description: Disease control rate (DCR) per modified RECIST 1.1 is defined as the percentage of participants with a best overall response of CR, PR or SD evaluated by blinded independent central review.
  CR was defined as the disappearance of all lesions except lymph node short axis < 10 mm; PR was defined as a ≥ 30% reduction in sum of diameters in target lesions. Confirmation of CR or PR was not required. SD was defined as neither sufficient shrinkage of target lesions to qualify for CR or PR nor sufficient increase to qualify for PD with ≥ 84 days elapsed after randomization.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 50.0 [44.73 to 55.27] | 56.6 [51.43 to 61.87]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.11, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.94 to 1.75] — [estimate comment as in outcome 11, analysis 1]

19. Secondary Outcome: Phase 3: Objective Response Rate Assessed Using Modified irRC-RECIST (iORR)
Description: Objective response rate per modified irRC-RECIST is defined as the percentage of participants with a best overall response of iCR or partial response assessed using modified irRC-RECIST (iPR) evaluated by blinded independent central review.
  iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment at least 4 weeks from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  iPR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation.
  Modifications to the irRC-RECIST 1.1 included an increase in the total number of target lesions and new measurable lesions to 10 with a maximum of 5 target lesions per organ, and target lesions must be measurable by CT or MRI only.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 39.9 [34.72 to 45.04] | 49.1 [43.87 to 54.40]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.020, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.06 to 1.96] — [estimate comment as in outcome 11, analysis 1]

20. Secondary Outcome: Phase 3: Best Overall Response Assessed Using Modified irRC-RECIST
Description: BOR is defined as the best overall visit response in the following order: iCR, iPR, stable disease per modified irRC-RECIST (iSD), iPD, or UE per modified irRC-RECIST (iUE), evaluated by BICR.
  iCR: Disappearance of all lesions confirmed by consecutive assessment ≥ 4 weeks from the date first documented. Reduction of any pathological lymph node to <10 mm.
  iPR: Decrease in tumor burden ≥ 30% relative to baseline confirmed ≥ 4 weeks after first documentation.
  iPD: Increase in tumor burden ≥ 20 % and at least 5 mm absolute increase relative to nadir confirmed ≥ 4 weeks from initial detection.
  iSD: Neither sufficient shrinkage to qualify for iCR or iPR nor sufficient increase to qualify for iPD and ≥ 84 days from randomization.
  Missing: No postbaseline assessment, or assessments after start of first subsequent anticancer therapy, including complete or partial removal/reduction of any target lesion which contained melanoma on pathology evaluation or pathology results were unknown.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
Participants
  Complete response (iCR) | 28 | 50
  Partial response (iPR) | 110 | 120
  Stable disease (iSD) | 57 | 51
  Progressive disease (iPD) | 56 | 65
  Unevaluable (iUE) | 69 | 30
  Missing | 26 | 30

21. Secondary Outcome: Phase 3: Durable Response Rate Assessed Using Modified irRC-RECIST (iDRR)
Description: Durable response rate per modified irRC-RECIST is defined as the percentage of participants with a best overall response of iCR or iPR per modified irRC-RECIST evaluated by blinded independent central review with a duration of response ≥ 6 months.
  iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment at least 4 weeks from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  iPR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 34.4 [29.39 to 39.40] | 45.7 [40.42 to 50.91]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.004, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.16 to 2.17] — [estimate comment as in outcome 11, analysis 1]

22. Secondary Outcome: Phase 3: Duration of Response Assessed Using Modified irRC-RECIST (iDOR)
Description: Duration of response per modified irRC-RECIST is defined as the time from the date of an initial response of iCR or iPR that was subsequently confirmed to the earlier of iPD per modified irRC-RECIST evaluated by blinded independent central review, or death. Participants who had not ended their response at the time of analysis were censored at their last evaluable tumor assessment date before the start of the first subsequent anticancer therapy.
  iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment at least 4 weeks from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  iPR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation.
Time Frame: as for outcome 12
Population: Participants randomized in Phase 3 with a iCR or iPR per modified irRC-RECIST.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 138 | 170
months | NA [NA to NA] — Could not be estimated due to the low number of events | 43.7 [34.53 to 43.73]

23. Secondary Outcome: Phase 3: Disease Control Rate Assessed Using Modified irRC-RECIST (iDCR)
Description: Disease control rate per modified irRC-RECIST is defined as the percentage of participants with a best overall response of iCR, iCR, or iSD assessed using modified irRC-RECIST evaluated by blinded independent central review.
  iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment at least 4 weeks from the date first documented. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  iPR: Decrease in tumor burden ≥ 30% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation.
  iSD: Neither sufficient shrinkage to qualify for iCR or iPR nor sufficient increase to qualify for iPD with ≥ 84 days elapsed after randomization.
Time Frame: as for outcome 11
Population: All participants randomized in Phase 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 346 | 346
percentage of participants | 56.4 [51.13 to 61.58] | 63.9 [58.81 to 68.93]
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Test type: Other; p = 0.058, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.99 to 1.85] — [estimate comment as in outcome 11, analysis 1]

24. Secondary Outcome: Phase 3: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Core Module (EORTC QLQ-C30) Global Health Status (GHS)/Quality of Life (QOL) Score
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status/quality of life scale, 5 functional scales, and 9 symptom scales/items.
  The global health/QoL scale consists of 2 questions that ask participants to rate their overall health and overall quality of life during the past week on a scale from 1 (very poor) to 7 (excellent). The GHS/QoL subscale score was derived as the mean of each score then transformed to a scale from 0 to 100 where higher scores represent a better health status and a positive change from baseline indicates improvement.
  The overall change from baseline (calculated from all on-treatment visits) was calculated using a restricted maximum likelihood-based mixed model for repeated measures (MMRM) (see model details in statistical analysis section).
Time Frame: Baseline and day 1 of weeks 3, 6, 9, 12, then every 6 weeks until end of study treatment; median (range) duration of treatment was 39.0 (0.1, 107.3) weeks in Placebo + Pembrolizumab and 54.1 (0.1, 109.6) weeks in Talimogene Laherparepvec + Pembrolizumab.
Population: Participants randomized in Phase 3 who received at least one dose of study therapy and had both a baseline and at least one on-treatment assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 329 | 328
score on a scale | -0.20 (1.02) | -0.02 (1.02)
Statistical Analysis 1: Comparison: Phase 3: Placebo + Pembrolizumab vs Phase 3: Talimogene Laherparepvec + Pembrolizumab; Mixed Model for Repeated Measures include the fixed and categorical effects of treatment, visit and treatment-by-visit interaction, the fixed and continuous covariates of baseline HRQL score, randomization stratification factors (stage of disease and prior BRAF inhibitor therapy per IVRS) and baseline PD-L1 status (positive and not positive). Random subject effect was modeled using within subject-error correlation structure; Test type: Other; p = 0.84, Mixed Model for Repeated Measures; Difference = 0.19, 95% CI 2-sided [-1.67 to 2.05], Standard Error of Mean 0.95

25. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial subject, including worsening of a pre-existing medical condition. The event does not necessarily have a causal relationship with study treatment. TEAEs include AEs from the first dose of study drug to 30 days after the last dose.
  A serious adverse event (SAE) is an AE that met at least 1 of the following criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. Treatment-emergent SAEs are any SAE occurring from first dose of study drug through 90 days after the last dose or 30 days after the last dose if new anticancer therapy was started, whichever was earlier.
  AEs were graded for severity using CTCAE version 4.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening; Grade 5 = Fatal.
Time Frame: From first dose to 30 days after last dose (90 days for SAEs); median (range) duration was 48 (5.1, 110.1) weeks in Phase 1b, 39 (0.1, 107.3) weeks in Placebo + Pembrolizumab and 56 (0.1, 109.6) weeks in Phase 3 Talimogene Laherparepvec + Pembrolizumab.
Population: All participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab. One participant who was randomized in Phase 3 to receive placebo received talimogene laherparepvec; thus, the Safety Analysis Set consisted of 344 participants in the Talimogene Laherparepvec + Pembrolizumab group and 344 participants in the Placebo + Pembrolizumab group.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 21 | 344 | 344
Participants
  Any treatment-emergent adverse events | 21 | 331 | 338
  Grade ≥ 2 | 20 | 279 | 306
  Grade ≥ 3 | 13 | 151 | 161
  Grade ≥ 4 | 2 | 29 | 33
  Serious adverse events | 8 | 141 | 154
  Leading to discontinuation of talimogene laherparepvec/Placebo | 0 | 24 | 26
  Leading to discontinuation of pembrolizumab | 2 | 41 | 43
  Fatal adverse events | 1 | 42 | 45

ADVERSE EVENTS:
Time Frame: All-cause mortality: From enrollment (Phase 1b) or randomization (Phase 3) to end of study, up to 75 months in Phase 1b and 58 months in Phase 3. SAEs: From first dose of study drug to 90 days after last dose or 30 days after last dose if new anticancer therapy was started. AEs: From first dose to 30 days after last dose; median (range) duration of exposure was 48 (5.1, 110) weeks in Phase 1b, 39 (0.1, 107) weeks in Placebo + Pembrolizumab and 56 (0.1, 110) weeks in T-VEC + Pembrolizumab arm.
Description: All-cause mortality is reported for all enrolled (Phase 1b) or randomized (Phase 3) participants.
  Adverse events are reported for all participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab.
  One participant who was randomized in Phase 3 to receive placebo received talimogene laherparepvec; thus, the Safety Analysis Set consisted of 344 participants in the talimogene laherparepvec + pembrolizumab group and 344 participants in the placebo + pembrolizumab group.
Arm/Group | Phase 1b: Talimogene Laherparepvec + Pembrolizumab | Phase 3: Placebo + Pembrolizumab | Phase 3: Talimogene Laherparepvec + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/21 | 156/346 | 146/346
Serious Adverse Events (participants affected / at risk) | 8/21 | 141/344 | 154/344
Other Adverse Events (participants affected / at risk) | 21/21 | 305/344 | 317/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Talimogene Laherparepvec + Pembrolizumab (N=21) | Phase 3: Placebo + Pembrolizumab (N=344) | Phase 3: Talimogene Laherparepvec + Pembrolizumab (N=344)
Anaemia (Blood and lymphatic system disorders) | 0 | 8 | 9
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Granulomatous lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3 | 4
Myocarditis (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Addison's disease (Endocrine disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0
Endocrine disorder (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 2 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 1 | 2
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 0 | 1
Retinal oedema (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 1
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Condition aggravated (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 2
Disease progression (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 3
General physical health deterioration (General disorders) | 1 | 2 | 1
Generalised oedema (General disorders) | 0 | 1 | 1
Inflammation (General disorders) | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 2 | 1
Pain (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 4 | 7
Sudden death (General disorders) | 0 | 1 | 1
Swelling (General disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 4 | 4
Chorioretinitis (Infections and infestations) | 0 | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2 | 2
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Lymph gland infection (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 4 | 3
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Scrotal abscess (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Ureteritis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 5
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 2
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 26 | 27
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 10 | 7
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0
Somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Axillary lymphadenectomy (Surgical and medical procedures) | 0 | 1 | 0
Arteritis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Labile blood pressure (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 2 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Talimogene Laherparepvec + Pembrolizumab (N=21) | Phase 3: Placebo + Pembrolizumab (N=344) | Phase 3: Talimogene Laherparepvec + Pembrolizumab (N=344)
Anaemia (Blood and lymphatic system disorders) | 2 | 26 | 33
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 20 | 22
Hypothyroidism (Endocrine disorders) | 6 | 49 | 48
Visual impairment (Eye disorders) | 2 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 24 | 23
Abdominal pain upper (Gastrointestinal disorders) | 2 | 12 | 7
Constipation (Gastrointestinal disorders) | 4 | 28 | 52
Diarrhoea (Gastrointestinal disorders) | 13 | 73 | 70
Dry mouth (Gastrointestinal disorders) | 1 | 19 | 14
Frequent bowel movements (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 61 | 92
Vomiting (Gastrointestinal disorders) | 7 | 29 | 56
Asthenia (General disorders) | 2 | 29 | 27
Chills (General disorders) | 8 | 17 | 73
Face oedema (General disorders) | 2 | 0 | 3
Fatigue (General disorders) | 15 | 94 | 137
Influenza like illness (General disorders) | 5 | 26 | 64
Injection site pain (General disorders) | 2 | 14 | 15
Injection site reaction (General disorders) | 2 | 3 | 10
Oedema peripheral (General disorders) | 5 | 22 | 27
Pain (General disorders) | 1 | 18 | 24
Pyrexia (General disorders) | 10 | 33 | 128
Cellulitis (Infections and infestations) | 2 | 9 | 14
Influenza (Infections and infestations) | 2 | 7 | 9
Nasopharyngitis (Infections and infestations) | 1 | 23 | 21
Oral herpes (Infections and infestations) | 2 | 16 | 15
Rhinitis (Infections and infestations) | 2 | 11 | 7
Upper respiratory tract infection (Infections and infestations) | 2 | 17 | 17
Urinary tract infection (Infections and infestations) | 1 | 17 | 22
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 2 | 5 | 9
Alanine aminotransferase increased (Investigations) | 3 | 23 | 26
Aspartate aminotransferase increased (Investigations) | 3 | 16 | 20
Blood alkaline phosphatase increased (Investigations) | 2 | 7 | 15
Blood iron decreased (Investigations) | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 26 | 43
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 11 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 66 | 82
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 30 | 35
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 16 | 33
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 21 | 29
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1
Headache (Nervous system disorders) | 9 | 44 | 62
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 4
Paraesthesia (Nervous system disorders) | 2 | 6 | 13
Anxiety (Psychiatric disorders) | 2 | 7 | 11
Insomnia (Psychiatric disorders) | 3 | 27 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 44 | 58
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 24 | 23
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 18
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 10
Erythema (Skin and subcutaneous tissue disorders) | 2 | 15 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 55 | 61
Rash (Skin and subcutaneous tissue disorders) | 9 | 42 | 61
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 17 | 20
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 11
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Vitiligo (Skin and subcutaneous tissue disorders) | 5 | 32 | 44
Hypertension (Vascular disorders) | 1 | 22 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT02263508/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT02263508/SAP_001.pdf